CLINICAL TRIAL: NCT03349450
Title: Phase 2 Study of an Immune Therapy, DPX-Survivac With Low Dose Cyclophosphamide Administered With Pembrolizumab in Patients With Persistent or Recurrent/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: DPX-Survivac and Checkpoint Inhibitor in DLBCL
Acronym: SPiReL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0891
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-07

CONDITIONS: Adult Diffuse Large Cell Lymphoma; Recurrent; Adult Refractory Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma; DLBCL; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Cyclophosphamide; Pembrolizumab; Immunosuppressive Agents; Immunologic Factors; Physiological Effects of Drugs; Antirheumatic Agents; Antineoplastic Agents, Alkylating; Alkylating Agents; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Myeloablative Agonists; Canada; Ontario; Diffuse Large B Cell Lymphoma; refractory; relapsed; checkpoint inhibitor; vaccine; DPX-Survivac; Survivin; Immunotherapy; Transformed Lymphoma; Double Hit; Large Cell Lymphoma; Keytruda
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma; Lymphoma, B-Cell; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; Dendritic Cell Sarcoma, Interdigitating | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm-Investigational (Experimental): DPX-Survivac Priming dose of 0.5ml. DPX-Survivac Booster dose of 0.1ml.
  Pembrolizumab 200mg Intravenously.
  Cyclophosphamide 50mg Twice daily orally.
  Interventions: Biological: DPX-Survivac; Biological: Pembrolizumab; Drug: Cyclophosphamide 50mg

INTERVENTIONS:
Biological: DPX-Survivac — DPX-Survivac Priming dose of 0.5ml on Study days 7 and 28. DPX-Survivac Booster dose of 0.1ml on Study days 84, 140, 196, 252, 308, and 364.
Biological: Pembrolizumab — Pembrolizumab 200mg administered intravenously every 3 weeks, commencing on study day 7 to a total of 18 infusions
Drug: Cyclophosphamide 50mg — Cyclophosphamide 50mg twice daily by mouth, administered 7 days on / 7 days off, stating at study day 0, until study day 384

SUMMARY:
This is a Phase 2 non-randomized, open label, uncontrolled, efficacy and safety study. Study participants will receive two priming doses of 0.5mL of DPX-Survivac 21 days apart and up to six 0.1ml maintenance injections every two months with low dose metronomic oral cyclophosphamide (50 mg BID) for one year or until disease progression, whichever occurs first.

Pembrolizumab 200 mg will be administered every 3 weeks for up to one year or until disease progression, whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase 2, non-randomized, open-label, uncontrolled, efficacy and safety trial.

Participants will receive 2 priming injections (0.5ml) of DPX-Survivac 3 weeks apart on Study Days 7 and 28. In addition, up to 6 maintenance injections (0.1ml) over the course of the study occurring on Study Days 84, 140, 196, 252, 308, and 364. All injections will be given under the skin of the upper thigh.

Participants will receive metronomic oral cyclophosphamide (50mg BID; 7 days on / 7 days off) for study period.

Pembrolizumab 200mg will be administered intravenously every 3 weeks, commencing on study day 7, to a total of 18 infusions.

If a participant is removed from the trial prior to the completion of at least 4 doses of Pembrolizumab and 3 injections of DPX-Survivac, that particiapnt may be replaced to determine the efficacy of treatment in a minimum of 16 participants.

DPX-Survivac injection sites will be evaluated throughout the study and if evidence of significant reaction, an Injection site reaction biopsy will be sought.

During the course of the study, blood will be drawn to evaluate immune cells and the effect that DPX Survivac will have on the participants immune system. During all treatment cycles a physical exam and questions about the participants general health will be performed.

Participants will undergo "re-staging" to assess the status of their disease at approximately study day 70 (if there is evidence of Grade 2 or greater injection site reaction or ulceration evident on study day 49) or routinely at approximately study day 91, and again at end of study or study withdrawal for all participants.

A follow-up tumour biopsy will be requested between study day 77-83 for participants with any grade 2 or greater Injection site reaction or ulceration on SD49 or between SD98 and SD104 if no evidence of injection site reaction or ulceration.

Upon completion of study, participants will be monitored every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Male or female 18+ years of age on day of signing informed consent and of any racial or ethnic group
3. Has:

   A. histologically proven DLBCL with recurrence after first, second or tertiary treatment regimens for DLBCL or,

   B. evidence of transformed lymphoma with past history of indolent lymphoma with current biopsy showing DLBCL) or,

   C. double hit or high grade lymphomas, including Burkitts lymphoma and High Grade B-Cell lymphoma unclassifiable (with features intermediate between Burkitts and diffuse large B cell lymphoma)
4. Has had:

   A. recurrence requiring therapy at least 90 days post aggressive first line combination chemotherapy (e.g. RCHOP, Hyper-CVAD or other aggressive "curative" combination), autologous stem cell transplantation (ASCT), CART therapy, or aggressive second line combination therapy or,

   B. partial response or measureable disease after first line therapy (who are not candidates for ASCT) or after second or third line therapy without disease progression or,

   C. recurrence any time after non-aggressive combination or single agent therapy with or without Rituximab (i.e. CVP, CHL or, VP16) for first, second or third line disease or,

   D. for subjects with transformed lymphoma, a treatment for indolent lymphoma within the last 2 years
5. Have at least one measurable site of disease based on Cheson Criteria using standard CT imaging.
6. Be willing to provide tissue from a newly obtained (up to 3 months + 7 days prior to Study Day 0) biopsy of a tumour lesion. If this is not available, the patient must be willing to undergo a core biopsy prior to starting treatment. They must also be willing to provide an on-treatment biopsy.
7. Have a performance status of 0-1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 2, within 48 hours prior to receiving the first dose of study medication (SD0). Patients with abnormal liver enzymes of up to 5 times the upper limit of normal and/or reduced GFR of 50-100% normal range can be considered for enrolment if the alteration is due to lymphoma.
9. Previous localized surgery, radiotherapy, chemotherapy, and immunotherapy more than 21 days prior to SD0. Cyclophosphamide, up to 100 mg/day, may be administered until SD-1 for subjects already receiving as a single agent therapy.
10. A life expectancy > 6 months.
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 48 hours prior to receiving the first dose of study medication (SD0). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through to 120 days from the last dose of study medication.
14. Ability to comply with protocol requirements.

Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 21 days of the first dose of treatment (SD0).
2. Patients eligible for possible curative therapies such as ASCT.
3. LDH greater than 5 times the upper limit of normal.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 35 days prior to the first dose of trial treatment (SD0), except that used as pre-medication for chemotherapy or contrast-enhanced studies are eligible. Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<10 mg daily).
5. Has had previous allogeneic stem cell transplant
6. Has known active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 21 days prior to SD0 or who has not recovered (i.e., ≤ Grade 1) from adverse events due to agents administered more than 21 days earlier.
9. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 21 days prior to SD0. Subjects must have recovered from all acute toxicities from prior treatments; peripheral neuropathy must be ≤ grade 2.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include in situ cervical cancer, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided; they are stable (without evidence of progression by imaging) for at least four weeks prior to the first dose of trial treatment; and any neurologic symptoms have returned to baseline; have no evidence of new or enlarging brain metastases; and are not using steroids for at least 35 days prior to trial treatment.
12. Progressive CNS lymphoma requiring treatment within 35 days prior to SD0.
13. Has history of active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has known history of, or any evidence of active, non-infectious pneumonitis.
15. Thyroiditis within the past 5 years.
16. Has an active infection requiring systemic therapy. Subjects completing a course of antibiotic for acute infection 7 days prior to SD0 and who do not experience a recurrence of symptoms or fever are eligible.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with screening visit to 120 days after last dose of study medication.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
22. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Evidence of Hepatitis B surface antigen without transaminitis is allowed provided patient is treated with anti-viral therapy (Heptavir or Tenofovir).
23. Patients who have received prior survivin based vaccines.
24. Acute or chronic skin disorders that will interfere with subcutaneous injection of the DPX-Survivac or subsequent assessment of potential skin reactions.
25. Serious intercurrent chronic or acute illness, such as cardiac disease (New York Heart Association class III or IV), hepatic disease, or other illness considered by the investigator as an unwarranted high risk for an investigational product.
26. Allergies to any vaccine, that after discussion with the medical monitor are serious enough to warrant exclusion from this study.
27. Received a live vaccine within 30 days of planned start of study therapy. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
To document the objective response rate using modified Cheson criteria to treatment with DPX-Survivac and low dose cyclophosphamide administered together with Pembrolizumab in participants with recurrent, survivin-expressing B cell lymphomas | 1 Year

SECONDARY OUTCOMES:
To document changes in tumour volume using waterfall analyses | 1 Year
  Tumor volume measurements will be obtained at multiple time points by adding the volumes of the perpendicular measurements for up to 6 target lesions
To document the toxicity profile | 1 Year
  Number of participants with abnormal laboratory values and/or adverse events related to treatment will be assessed.
To document duration of response using modified Cheson criteria. | 2 Years
  Completing response assessment post radiology
To document time to next treatment | 2 Years
  time lapse between current and next treatment

OTHER OUTCOMES:
Exploratory Outcome 1 | 1 year
  (1) To document the changes in circulating T cell immune responses to survivin and relationship to peripheral B cell numbers
Exploratory Outcome 2 | 1 year
  To document changes in T cell and T cell subset infiltration and gene expression pathways in treatment compared to pre-treatment tumour biopsies
Exploratory Outcome 3 | 1 year
  To assess potential biomarkers of immune and clinical response from pre-treatment and on-treatment tumor biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Neil L Berinstein, MD, Principal Investigator — Sunnybrook Research Institute
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre - Alberta Health Services, Calgary, Alberta
  - Nova Scotia Health Authority: Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
For original data, contact SPiReL@sunnybrook.ca. Individual patient data will not be de-identified, however, data can be shared for a period of up to 5 years after trial closure with formal Confidentiality and Data Transfer agreements in place as appropriate.
  A data dictionary will not be shared, but the study protocol can be found on ClinicalTrials.gov with trial #NCT03349450 and the Statistical Analysis Plan can be made available with publication.
Supporting Information: Study Protocol
Time Frame: Up to 5 years after the closure of the trial

REFERENCES:
- [Result] Amitai I, Roos K, Rashedi I, Jiang Y, Mangoff K, Klein G, Forward N, Stewart D, Laneuville P, Bence-Bruckler I, Mangel J, Tomlinson G, Berinstein NL. PD-L1 expression predicts efficacy in the phase II SPiReL trial with MVP-S, pembrolizumab, and low-dose CPA in R/R DLBCL. Eur J Haematol. 2023 Aug;111(2):191-200. doi: 10.1111/ejh.13982. Epub 2023 May 8. PMID 37157906
- [Derived] Pandey A, Roos K, Jiang Y, Mangoff K, Klein G, Forward N, Stewart D, Laneuville P, Bence-Bruckler I, Mangel J, Tomlinson G, Berinstein NL. Characteristics of relapsed/refractory diffuse large B-cell lymphoma patients with durable responses to maveropepimut-S, pembrolizumab, and cyclophosphamide: Long-term follow-up from the SPiReL trial. EJHaem. 2024 Dec 12;6(1):e1062. doi: 10.1002/jha2.1062. eCollection 2025 Feb. PMID 39866944

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03349450/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03349450/SAP_001.pdf